CLINICAL TRIAL: NCT03229746
Title: Reposition of Second Line Treatment in Chronic Immune Thrombocytopenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada E. M. Abdallah, Principal investegator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17200058
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Hydroxychloroquine; Vincristine; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- hydroxychloroquine group (Experimental): hydroxychloroquine tablets 200mg ,two times/day for at least 6 month
  Interventions: Drug: Hydroxychloroquine
- vincristine group (Active Comparator): vincristine ampoule , 1mg/ week, I.v drep over 2 hours for 4 weeks
  Interventions: Drug: vincristine
- azathioprine group (Active Comparator): azathioprine tablet 50mg, dose 100-150 mg daily for 6 month
  Interventions: Drug: azathioprine

INTERVENTIONS:
Drug: Hydroxychloroquine — 200mg twice daily orally for at least 12 weeks
  Arms: hydroxychloroquine group
Drug: vincristine — 1mg intravenous weekly for 4 weeks
  Arms: vincristine group
Drug: azathioprine — dose 100mg daily for at least 3 weeks
  Other Names: imuran
  Arms: azathioprine group

SUMMARY:
Hydroxychloroquine has been reported to have a clinically significant effect on the platelet count in systemic lupus thrombocytopenia. Its action may be due to its immune modulator effect. Immune thrombocytopenia (ITP) is known as an immune-mediated acquired disease characterized by transient or persistent decrease of the platelet count. However, refractory ITP is lacking of effective treatments and the efficacy of decitabine in ITP remains poorly understood. Data from this study may provide some idea of Hydroxychloroquine in the treatment of ITP in comparison to other lines of treatment as detected by the standardized definitions.

DETAILED DESCRIPTION:
This study will include patients with chronic ITP attending the out patients clinic of Clinical Hematology Unit of Internal Medicine Department of Assiut university Hospital to evaluate the safety and efficacy of hydroxychloroquine in comparison to other lines of treatment as detected by the standardized definitions . Detect the predictors for chronic ITP especially anti-nuclear antibodies (ANA) role and the effect of the proposed drugs on the level of anti-platelet antibodies. Evaluation of the health-related quality of life after treatments to answer this question; Is the most effective drug is linked to the best quality of life.

ELIGIBILITY:
Inclusion Criteria:

* We will recruit patients with primary chronic ITP patients with ITP lasting for more than 12 months which is proved to be refractory to the standard first line treatment or need to treatment(s) (including, but not limited to, low dose of corticosteroids) to minimize the risk of clinically significant bleeding.
* Subject or their guardian has signed and dated a written informed consent.
* Subject experienced no toxicity or known contraindication to any line of treatments.

Exclusion Criteria:

* pregnancy.
* liver and kidney function impairment.
* hepatitis c virus(HCV), human immunodeficiency virus (HIV), hepatitis B virus infection.
* patients with systemic lupus erythematosus and/or antiphospholipid syndrome
* lymphoproliferative disorders.
* an active malignancy
* an arterial or venous thrombosis
* Grade III-IV cardiovascular disease .
* Recent history of alcohol/drug abuse.
* Subjects recently treated with drugs that affect platelet function (including but not limited to aspirin, clopidogrel and/or NSAIDs) or anti-coagulants for > 3 consecutive days within 2 weeks of the study start and until the end of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Platelet count | Follow up untill response or death from any cause up to six months
  to detect response as the standard definition
side effects | Up to six months
  any complication for any line of treatments line

SECONDARY OUTCOMES:
anti- nuclear antibodies role | before enrollment
  Detecting the predictors for chronic ITP especially ANA role
Anti-platelets antibodies role | after6 months
  Evaluation of the effect of the proposed drugs on the level of anti-platelet antibodies .
Health quality life | after 6 months of treatment
  The Arabic version of the 36-Item Short Form Survey Instrument (SF-36) questionnaire will be administered to all patients before & after treatment.
  This questionnaire is a validated one which assesses general health functioning .

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park YH, Yi HG, Lee MH, Kim CS, Lim JH. Clinical efficacy and tolerability of vincristine in splenectomized patients with refractory or relapsed immune thrombocytopenia: a retrospective single-center study. Int J Hematol. 2016 Feb;103(2):180-8. doi: 10.1007/s12185-015-1903-0. Epub 2015 Nov 20. PMID 26588926
- [Background] Poudyal BS, Sapkota B, Shrestha GS, Thapalia S, Gyawali B, Tuladhar S. Safety and Efficacy of Azathioprine as a Second Line Therapy for Primary Immune Thrombocytopenic Purpura. JNMA J Nepal Med Assoc. 2016 Jul-Sep;55(203):16-21. PMID 27935917
- [Background] Cooper N. State of the art - how I manage immune thrombocytopenia. Br J Haematol. 2017 Apr;177(1):39-54. doi: 10.1111/bjh.14515. Epub 2017 Mar 10. PMID 28295192
- [Background] Michel M. Immune thrombocytopenic purpura: epidemiology and implications for patients. Eur J Haematol Suppl. 2009 Mar;(71):3-7. doi: 10.1111/j.1600-0609.2008.01206.x. PMID 19200301
- [Result] Khellaf M, Chabrol A, Mahevas M, Roudot-Thoraval F, Limal N, Languille L, Bierling P, Michel M, Godeau B. Hydroxychloroquine is a good second-line treatment for adults with immune thrombocytopenia and positive antinuclear antibodies. Am J Hematol. 2014 Feb;89(2):194-8. doi: 10.1002/ajh.23609. Epub 2013 Nov 20. PMID 24254965